CLINICAL TRIAL: NCT06740968
Title: Improving Neural Oscillation and Synchrony Between Motor and Auditory Regions in Stuttering Using Personalized Transcranial Alternating Current Stimulation (tACS)
Brief Title: Transcranial Alternating Current Stimulation (tACS) in Stuttering
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Soo-Eun Chang, Associate Professor of Psychiatry, University of Michigan
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HUM00211167
Record Dates: First submitted 2024-12-14; First posted 2024-12-18 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Stuttering, Adult; Stuttering, Childhood; Stuttering, Developmental
Keywords: tACS; Magnetic resonance imaging; Electroencephalogram; Auditory perturbation; Neural oscillations; Brain stimulation
MeSH Terms: conditions — Stuttering | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: Participants will all receive the same treatments, however, visits 3 through 5 will have order of conditions (types of stimulation) randomized.
Masking Description: Please note that because the most logical interventional study model is a single arm study the study team can't select a masking option. Please note that Participants, Investigators, and Outcomes Assessors will be blinded to active vs. sham stimulation (with the exception of one study investigator that pre-configures the randomization schedule, and this person will not be involved in any assessments/outcomes).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- transcranial alternating current stimulation (tACS) (Experimental): Participants will receive 3 sessions of tACS. Each session can be active or sham. The stimulation parameters regarding the active and sham will not be disclosed at this time to maintain blind to participants. At the end of the trial the study will be updated to list these.
  Interventions: Device: transcranial alternating current stimulation (tACS)

INTERVENTIONS:
Device: transcranial alternating current stimulation (tACS) — During each of the 3 stimulation visits, participants will be seated in a comfortable position and a cap will be placed on participant's head similar to a swimming cap. Small electrodes will be placed near the surface of the scalp at certain regions of interest, and a weak electrical current will be passed through the electrodes into speech related brain areas for 20 minutes. The study team will not use current strengths exceeding 2 milliamps (mA).

SUMMARY:
The purpose of this study is to investigate how mild, noninvasive electrical brain stimulation affects speech relevant brain areas, which may in turn affect speech fluency and speaking-related brain activity in people that stutter. The long-term goal of this study is to test the therapeutic potential of transcranial alternating current stimulation (tACS) for the treatment of stuttering.

The study team hypothesizes that if stuttering involves impaired initiation of motor programs, delta-tuned tACS will strengthen communication between brain regions and decrease stuttering. Therefore, delta-tuned sensorimotor tACS will be paired with fluency-induced speech (choral reading), which is hypothesized to decrease stuttering via improved auditory motor integration.

DETAILED DESCRIPTION:
Participants will have screening and baseline visits that include a variety of tests and procedures (i.e. standardized tests of speech, language, hearing test, music training questionnaire, working memory tests, and speech sample to characterize stuttering, magnetic resonance imaging (MRI) and electroencephalography (EEG)). Following these, participants will have 3 sessions (active and sham conditions) and then a one month follow-up phone or video call.

Of note, there will be an embedded pilot study to refine the experimental protocol in terms of practicality and feasibility and these participants will not be included in this registration. The only purpose of this embedded study is to refine the protocol and it does not have any health or behavioral outcomes.

ELIGIBILITY:
Inclusion Criteria for stutterers:

* Have normal language, hearing, and cognition
* Speak English as the primary language
* Currently stutter
* Score (per protocol) a certain value on the Stuttering Severity Instrument (SSI-4).
* Have not received any treatment for stuttering within the past year

Exclusion Criteria for stutterers:

* History of seizures
* Major medical or neurological illness (e.g., stroke, serious head trauma, brain infection, Parkinson's disease, etc.)
* History of closed head injury with loss of consciousness (e.g., concussion)
* Metal or electronic implants such as cochlear implants and pacemakers anywhere in the body
* Braids or other hair styling that prevents direct access to the scalp (if removal not possible)
* Currently pregnant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-08-05 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Change in Phase Synchronization | Baseline (pre-tACS), approximately 3 hours (post-tACS) (visits 3-5)
  The study will compare EEG data recorded before and after stimulation to determine if tACS contributed to any changes. This will be measured by Phase Locking Value (PLV; measured from 0 to 1) between the two regions targeted by stimulation calculated as [pre(active-sham)] - [post(active-sham)] at each tACS visit.

SECONDARY OUTCOMES:
Percentage of stuttered syllables produced during speech sample | Baseline (before tACS), approximately 3 hours (post-tACS) (visits 3-5)
  The study will calculate the percentage of stuttered syllables (out of total syllables) in a speech sample. Decreased stuttered syllables represents better outcomes (greater reduction in stuttering).

OTHER OUTCOMES:
Percent change in perturbation response | Baseline (before tACS), approximately 3 hours (post-tACS) (visits 3-5)
  The study will compare the perturbation task from before and after tACS. This is measured by the percent change in perturbation response.
Change in Phase Amplitude Coupling | Baseline (before tACS), approximately 3 hours (post-tACS) (visits 3-5)
  The study will compare EEG data recorded before and after stimulation to determine if tACS contributed to any changes. Phase Amplitude Coupling (PAC) will be calculated within and between the two regions targeted by stimulation calculated as [pre(active-sham)] - [post(active-sham)] at each tACS visit.

CONTACTS AND LOCATIONS:
Overall Officials: Soo-Eun Chang, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No